CLINICAL TRIAL: NCT01768728
Title: A Randomized Controlled Trial of Acute Surgical Trauma and Stress Response of Laparoscopic Versus Open Left Hemihepatectomy for Liver Benign Lesions
Brief Title: Laparoscopic Versus Open Left Hemihepatectomy for Liver Benign Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiujun Cai, Executive Vice-President, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SRRSH20121225-1
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Benign Lesions in Left Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Laparoscopic left hemihepatectomy group (Active Comparator): Group of patients that are operated with laparoscopic left hemihepatectomy
  Interventions: Procedure: Laparoscopic left hemihepatectomy
- Open left hemihepatectomy (Active Comparator): Group of patients operated with open left hemihepatectomy
  Interventions: Procedure: Open left hemihepatectomy

INTERVENTIONS:
Procedure: Laparoscopic left hemihepatectomy — participants will be performed with laparoscopic left hepatectomy using laparoscopic instruments
  Other Names: Laparoscopic left hepatectomy
  Arms: Laparoscopic left hemihepatectomy group
Procedure: Open left hemihepatectomy — participants will be performed with traditional open left hepatectomy using laparotomic instruments
  Other Names: Open left hepatectomy
  Arms: Open left hemihepatectomy

SUMMARY:
The purpose of this study is to investigate the influence of the laparoscopic and open left hemihepatectomy on acute surgical trauma and stress response.

ELIGIBILITY:
Inclusion Criteria:

* patient with benign lesions who requires left hemihepatectomy
* Child-Pugh classification of A to B
* American Society Of Anesthesiologists (ASA) grading of I to III
* a body mass index of between 18 and 35
* willingness to participate in the study
* able to understand the nature of the study and what will be required of them

Exclusion Criteria:

* pregnant or lactating women
* unwillingness to participate
* Child-Pugh classification of C
* ASA grading of IV to V
* with condition of acute inflammatory,fever or diabetes mellitus
* with autoimmune disease or immunodeficiency
* taking drugs that affect the immune system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Plasma C-reactive protein (CRP) level | up to 7 days
  CRP will be tested before operation, 3,12,24 hours and 3,5,7 days after operation

SECONDARY OUTCOMES:
Inflammatory response markers including interleukin-6, interleukin-10 concentrations and tumor necrosis factor α level in serum | up to 7 days
  interleukin-6 and interleukin-10 will be tested before operation, 3,12,24 hours and 3,5,7 days after operation
Oxidative stress status including plasma malondialdehyde level and total antioxidant capacity | up to 7 days
  plasma malondialdehyde level and total antioxidant capacity will be tested before operation, 3,12,24 hours and 3,5,7 days after operation
Immune status including white blood cell count and human leukocyte antigen DR (HLA-DR) expression | up to 7 days
  white blood cell count and human leukocyte antigen DR (HLA-DR) expression will be tested before operation, 3,12,24 hours and 3,5,7 days after operation
Status of insulin resistant | up to 7 days
  Status of insulin resistant will be tested before operation, 3,12,24 hours and 3,5,7 days after operation
Systemic inflammatory response syndrome | up to 7 days
Status of hepatic cell apoptosis including hematoxylin and eosin (HE) staining, immunohistochemistry staining and caspase-3 expression | 24 hours
Time to functional recovery | Participants will be followed for the duration of hospital stay, an expected average of 7 days
Postoperative hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 8 days
Morbidity and mortality | up to 1 month
Quality of life | up to 1 month
Intraoperative parameters including operation time, pneumoperitoneum time, liver resection time, intraoperative estimated blood loss,transfusion | participants will be followed for the duration of operation, an expected average of 120 minutes

OTHER OUTCOMES:
Hospital costs | Participants will be followed for the duration of hospital stay, an expected average of 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China